CLINICAL TRIAL: NCT06644560
Title: A Nutrition and Exercise Prehabilitation Intervention on Inflammatory Biomarkers in American Indian Cancer Patients
Brief Title: A Nutrition & Exercise Prehabilitation Intervention on Inflammatory Biomarkers in AI Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004848; K08CA276137 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Obesity
Keywords: Obesity-related cancer; Nutrition and Exercise Prehabilitation Intervention; Inflammatory biomarkers
MeSH Terms: conditions — Neoplasms; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation Intervention (Experimental): This is a single-arm, pre-post, window of opportunity trial. The tailored prehab program will be implemented for AI cancer patients preparing for cancer surgery for a 3-week duration in the preoperative window of opportunity. The prehab intervention is designed to modify inﬂammatory biomarkers in paired pre/post-intervention blood and tissue samples. 30 individuals who are 18-80 years old with a diagnosis of obesity-related solid tumor cancer, scheduled at least 3 weeks out from cancer surgery who are receiving care at SCAHC will be recruited over the duration of the study. Blood samples will be collected before and after the prehab, and inflammatory biomarkers will be measured in the paired pre/post blood sample. Unstained slides from the diagnostic biopsy and resected tumor specimen will be requested, and inflammatory biomarkers will be measured in the paired pre/post tissue sample.
  Interventions: Behavioral: Prehabilitation Intervention

INTERVENTIONS:
Behavioral: Prehabilitation Intervention — The intervention involves a 3-week prehabilitation program during the participant's preoperative window before cancer surgery. During the intervention, patients will be asked to consume 60 grams of walnuts daily, participate in two 60-minute individualized supervised physical activity training sessions per week, meet with a nutritionist for a 30-60 minute session, and conduct 30 minutes of independent walking per day. The participants will be given pre-portioned walnuts for daily consumption, a pedometer, and educational materials. The participants will track their completion of tasks with a daily log and the study coordinator will also track their attendance at scheduled nutrition and fitness sessions. In addition, the study coordinator will check-in with participants twice weekly and send text reminders about their required activities.
  Other Names: Prehab Intervention

SUMMARY:
The purpose of this study is to assess the feasibility of a prehab intervention among American Indian (AI) patients diagnosed with obesity-related cancer and measure inflammatory biomarkers to evaluate the preliminary impact of the trial intervention. The central hypothesis is that this community-informed prehab intervention will demonstrate feasibility, patient acceptability, and modulation of host and tumor-microenvironment inflammatory biomarkers.

Aim 1: Implement the prehab translational clinical trial for AI patients with obesity-related solid tumor cancer scheduled for surgery.

Aim 2 Measure host and tumor-microenvironment (TME) biomarkers using paired serum and tissue samples to compare baseline and post-intervention levels of expression. Serum markers include CRP, IL-6, IL-10, TNFa, IGF-1, VEGF, complete blood count (CBC) with differential, comprehensive metabolic panel (CMP), and prealbumin. Tissue markers include Ki67, insulin receptor, TNFa, NFKB, NOS2, and cleaved caspase 3.

Aim 3: (optional exploratory aim): Assess differential expression of inflammatory genes in the TME using tumor tissue samples to compare baseline and post-intervention levels of expression. This will be done with a panel that analyzes inflammatory genes only.

DETAILED DESCRIPTION:
The research entails a single-arm, pre-post, window-of-opportunity prehab intervention trial. The tailored prehab program will be implemented for cancer patients receiving care at San Carlos Apache Healthcare Corporation (SCAHC) who are preparing for cancer surgery for a 3-week duration in the preoperative window of opportunity. The prehab intervention is designed to modify inﬂammatory biomarkers in paired pre/post-intervention blood and tissue samples.

For the pilot intervention, 30 individuals who are 18-80 years old with a diagnosis of obesity-related solid tumor cancer, scheduled at least 3 weeks out from cancer surgery who receive care at SCAHC will be recruited over the duration of the study. Participants meeting criteria will be screened for eligibility. Those meeting eligibility criteria who are interested will be consented and enrolled. They will undergo baseline measurements that include medical/ family/cancer history and demographics, baseline anthropometric measures (blood pressure, weight, height, and waist circumference), completion of diet/exercise and health behavior questionnaires, 6-minute walk test, sit-to- stand test and blood samples which will be run for inﬂammatory biomarkers. The consent will include permission to obtain the diagnostic biopsy tissue for the purposes of this research study to measure tissue biomarkers.

After baseline evaluation, patients will receive diet and exercise counseling prior to commencing the prehab program. They will receive general nutritional guidance on healthy eating, walking, and instructed on the methods of self-monitoring their activity levels (pedometer, daily log, checklists). They will participate in twice weekly 60-minute training sessions supervised by certiﬁed fitness trainers and perform 30 minutes of walking daily on their own. They will consume 60g of walnuts (1/2cup) which can be consumed raw or incorporated into meals and recipes of their choosing. Participants will return to the clinic after 3 weeks of the prehab program to repeat all baseline metrics and participate in an exit interview. Residual tissue from the surgical specimen after clinical assessments are completed will be used to measure post-intervention biomarker expression.

Paired pre/post-intervention blood and tissue samples will be stored and analyzed for biomarker expression at the University of Arizona Shared Resources. Analysis of the qualitative data from the exit interviews and the biospecimens will be conducted at the University of Arizona.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Clinical diagnosis of obesity-related solid tumor cancer: obesity-related solid tumor cancers include thyroid, breast, liver, gallbladder, gastric, pancreatic, colorectal, ovarian, uterine, kidney, esophageal cancers.
* Preoperative status with plan to undergo an operation to remove the tumor
* Scheduled at least 3 weeks out from the operation
* Receiving care at San Carlos Apache Healthcare Corporation (SCAHC)
* Must be having cancer surgery at San Carlos Apache Healthcare Corporation or Banner University Medical Center-Tucson

Exclusion Criteria:

* Current or planned receipt of chemotherapy during the preoperative study period
* Digestive tract disease that would restrict diet modifications
* Allergy to the foods intended for the nutrition intervention
* Uncontrolled cardiac disease or other contraindications to moderate-intensity exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient enrollment and retention: proportion of patients who initiate the intervention, provide pre-intervention measurements and return for post-intervention measurements | Baseline and post-intervention (an average of 5 weeks)
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring patient reported acceptability via patient enrollment and retention. Patient retention will be estimated as the proportion of patients who initiate the intervention, provide pre-intervention measurements and return for post-intervention measurements, with an exact 95% binomial confidence interval.
Adherence to study protocol: compliance with intervention foods (walnuts) | 3 weeks during participant's preoperative window
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring patient reported acceptability via compliance with intervention foods (walnuts). Compliance with intervention foods (walnuts) will be estimated as the number of daily packets eaten/number distributed, with an exact 95% binomial confidence interval.
Adherence to study protocol: compliance with exercise recommendations | 3 weeks during participant's preoperative window
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring patient reported acceptability via compliance with exercise recommendations. Compliance with exercise recommendations will be estimated as the increase in daily steps (as measured by pedometers) post- versus pre-intervention using a 95% confidence interval.
Assessing patient acceptability via exit interviews to solicit patient experience and feedback | 3 weeks during participant's post-intervention assessment
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring patient reported acceptability via exit interviews. The exit interviews will provide qualitative data for assessment. The interview transcriptions will be coded and themed. Themes will be vetted with SCAHC staff to ensure shared understanding of concepts and accurate representation of community perspective.
Comparison of pre/post-intervention 6 Minute Walk Test Scores to assess lifestyle behavioral change | Baseline and post-intervention assessment (an average of 3 weeks)
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring lifestyle behavioral changes via the 6 Minute Walk Test scores. The score of the 6MWT is the distance a patient walks in 6 minutes. Pre/post intervention performance changes on the 6MWT will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Comparison of pre/post-intervention sit-to-stand test scores to assess lifestyle behavioral change | Baseline and post-intervention assessment (an average of 3 weeks)
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring lifestyle behavioral changes via the sit-to-stand test scores. The sit-to-stand test score is the total number of stands within 30 seconds (more than halfway up at the end of 30 seconds counts as a full stand). Pre/post intervention performance changes on the sit-to-stand test will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Comparison of pre/post-intervention patient responses to the Dietary Screener Questionnaire | Baseline and post-intervention assessment (an average of 3 weeks)
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring lifestyle behavioral changes via comparing pre/post- intervention responses to the Dietary Screener Questionnaire. The Dietary Screener Questionnaire has 30 questions. There is a scoring algorithm that converts the responses to estimates of dietary intake of fruits and vegetables, dairy, added sugar, whole grain, fiber, and calcium. Changes between pre and post intervention will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Comparison of pre/post-intervention patient responses to the Arizona Activity Questionnaire | Baseline and post-intervention assessment (an average of 3 weeks)
  Primary endpoint: determining feasibility of the prehabilitation intervention by measuring lifestyle behavioral changes via comparing Arizona Activity Questionnaire. The Arizona Activity Questionnaire has 14 sections with 77 line items. There is a formula that converts the responses to estimates of total energy expenditure and physical activity energy expenditure. Changes between pre and post intervention will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Assessing biosample collection rates: percentage of patients completing blood and tissue sample collection | Baseline and post-intervention assessment (an average of 3 weeks)
  Primary endpoint: determining feasibility of the prehabilitation intervention by assessing percentage of patients who complete blood and tissue sample collections. Biosample collection rates (plasma and tissue) will be estimated as the proportion of patients who provide biospecimens at the pre- and post-intervention visits, with exact 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Assess stability of anthropometric measures: blood pressure | Baseline and post-intervention assessment (an average of 3 weeks)
  Blood pressure is measured in units of millimeters of mercury (mmHg). Pre/post intervention changes will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Assess stability of anthropometric measures: weight | Baseline and post-intervention assessment (an average of 3 weeks)
  Weight will be measured in kilograms. Pre/post intervention changes will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Assess stability of anthropometric measures: waist circumference | Baseline and post-intervention assessment (an average of 3 weeks)
  Waist circumference will be measured in centimeters. Pre/post intervention changes will be estimated using 95% confidence intervals, with transformation as needed to induce normality.
Assess changes between pre and post intervention levels of serum biomarkers. | Baseline and post-intervention assessment (an average of 3 weeks)
  Serum biomarkers [including CRP, IL-6, IL-10, TNFa, IGF-1, VEGF, complete blood count (CBC) with differential, comprehensive metabolic panel (CMP), and prealbumin] will be quantified with ELISA. Changes in serum biomarker levels will be estimated using 95% confidence intervals.
Assess changes between pre and post intervention levels of tissue biomarkers. | Baseline and post-intervention assessment (an average of 3 weeks)
  Tissue biomarkers [including Ki67, insulin receptor, TNFa, NFKB, NOS2, cleaved caspase 3] will be quantified with ELISA. Changes in tissue biomarker levels will be estimated using 95% confidence intervals.

OTHER OUTCOMES:
Assess differential expression of inflammatory genes in the tumor microenvironment | Baseline and post-intervention (an average of 3 weeks)
  For patients who agree to the optional exploratory aim, the existing diagnostic biopsy tissue and surgical specimen tissue can be additionally analyzed for gene expression data. Genes related to inflammation would be measured and no other genes would be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Erdrich, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No